CLINICAL TRIAL: NCT05994963
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, 2-PART CROSSOVER STUDY TO ASSESS THE RELATIVE BIOAVAILABILITY OF SISUNATOVIR FOLLOWING SINGLE ORAL DOSE OF DIFFERENT FORMULATIONS UNDER FED AND FASTED CONDITIONS IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Compare Different Preparations of Sisunatovir in Healthy Adult Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C5241013; 2023-505228-79-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — sisunatovir

STUDY DESIGN:
Intervention Model Description: Two Parts, Crossover study
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 Treatment A (Experimental): 4 capsules of sisunatovir in fasted state
  Interventions: Drug: sisunatovir
- Part 1 Treatment B (Experimental): 2 tablets of sisunatovir in fasted state
  Interventions: Drug: sisunatovir
- Part 1 Treatment C (Experimental): 2 tablets of sisunatovir with a high-fat meal
  Interventions: Drug: sisunatovir
- Part 2 Treatment B (Experimental): 2 tablets of sisunatovir in fasted sate
  Interventions: Drug: sisunatovir
- Part 2 Treatment D (Experimental): 2 tablets of sisunatovir with a low-fat meal
  Interventions: Drug: sisunatovir

INTERVENTIONS:
Drug: sisunatovir — Administered as either capsules in fasted state or tablet in fasted or fed state.
  Other Names: PF-07923568; RV521

SUMMARY:
The purpose of this study is to learn how different preparations of sisunatovir are taken up into the blood when taken on an empty stomach or with a meal in healthy adults.

This study has two Parts and is seeking participants who:

- are healthy males or females of 18 years of age or older.

Part 1:

All participants will receive treatments: A, B, and C. The participants will be assigned to take medicines A, B or C by chance, like drawing names out of a hat.

All treatments will be taken by mouth.

* Participants assigned to treatment A will take four capsules of sisunatovir on empty stomach.
* Participants assigned to treatment B will take two sisunatovir tablets on empty stomach.
* Participants assigned to treatment C will take two sisunatovir tablets with a high-fat meal.

Part 2:

All participants will receive treatments: B and D. The participants will be assigned to take medicines B and D by chance, like drawing names out of a hat.

All treatments will be taken by mouth.

* Participants assigned to treatment B will take two sisunatovir tablets on empty stomach.
* Participants assigned to treatment D will take two sisunatovir tablets with a low-fat meal.

The participants will be in the study clinic for 10 days in Part 1 and 7 days in Part 2, for:

* safety checks,
* sample collection for lab tests,
* understanding how different preparations of sisunatovir are taken up into the blood when taken on an empty stomach or with a meal.

All participants selected in the study will be required to go through a screening period up to 28 days. A screening period is the time during which a few participants are tested to see whether they are fit for the study. The participants can join the study only if they are tested be fit and are interested to take part in the study.

The participants will be allowed to go home on Day 10 during Part 1, and on Day 7 during Part 2. About 28 to 35 days after being sent home following the final treatment, the participant will be contacted for a follow up visit either in person or by telephone. This is to check up on how the participant is doing and to end the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 years of age or older, inclusive, at the time of signing of the informed consent document (ICD).

   • All fertile participants must agree to use a highly effective method of contraception.
2. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac evaluation.
3. Body mass index (BMI) of 18 to 32 kg/m2; and a total body weight >45 kg (100 lb).

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

   * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
   * History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
2. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
3. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention, with the exception of moderate/strong CYP3A inducers or time-dependent inhibitors which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention
4. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
5. A positive urine drug test, confirmed by a repeated test, if deemed necessary.
6. For participants <60 years: Screening supine BP ≥140 mm Hg (systolic) or

   * 90 mm Hg (diastolic), following at least 5 minutes of supine rest. For participants
   * 60 years old, a screening supine BP of ≥150/90 mm Hg may be used. If systolic BP is ≥ 140 or 150 mm Hg (based on age) or diastolic ≥90 mm Hg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
7. Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate- age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third- degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the uncorrected QT interval is >450 ms, this interval should be rate-corrected using the Fridericia method only and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
8. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * eGFR <60 mL/min/1.73m2 based on CKD-EPI equation; AST or ALT level ≥1.05× ULN;
   * GGT>1.05× ULN;
   * ALP >1.05× ULN;
   * Total bilirubin level ≥1.05× ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
9. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
10. History of sensitivity to sisunatovir or any of the formulation components.
11. Use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes/day or 2 chews of tobacco/day
12. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5241013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study had 2 parts: Part 1 and Part 2. Total enrolled participants were 25 (Part 1=14 and Part 2=11).
Pre-assignment Details: Sisunatovir 200 milligram (mg) single oral dose was administered as powder in capsule (PIC) or wet granulation tablet (WGT) under fasted condition, or as WGT with food. Study had 2 parts: 1 and 2. Part 1, treatments were: A= sisunatovir 200 mg PIC under fasted condition; B = sisunatovir 200 mg WGT under fasted condition; C= sisunatovir 200 mg WGT with a high-fat meal. Part 2, treatments were: B = sisunatovir 200 mg WGT under fasted condition; D= sisunatovir 200 mg WGT with a low-fat meal.
Groups:
- Part 1: Treatment A Then Treatment B Then Treatment C: Participants received treatment A on Day 1 of Period 1. Period 1 was followed by Period 2, where participants received treatment B on Day 1 of Period 2. Period 2 was followed by Period 3, where participants received treatment C on Day 1 of Period 3.
- Part 1: Treatment B Then Treatment A Then Treatment C: Participants received treatment B on Day 1 of Period 1. Period 1 was followed by Period 2, where participants received treatment A on Day 1 of Period 2. Period 2 was followed by Period 3, where participants received treatment C on Day 1 of Period 3.
- Part 2: Treatment B Then Treatment D: Participants received treatment B on Day 1 of Period 1. Period 1 was followed by Period 2, where participants received treatment D on Day 1 of Period 2.
- Part 2: Treatment D Then Treatment B: Participants received treatment D on Day 1 of Period 1. Period 1 was followed by Period 2, where participants received treatment B on Day 1 of Period 2.
Period: Part 1: Treatment Period 1
Arm/Group | Part 1: Treatment A Then Treatment B Then Treatment C | Part 1: Treatment B Then Treatment A Then Treatment C | Part 2: Treatment B Then Treatment D | Part 2: Treatment D Then Treatment B
Started | 7 | 7 | 0 | 0
Completed | 7 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1: Treatment Period 2
Arm/Group | Part 1: Treatment A Then Treatment B Then Treatment C | Part 1: Treatment B Then Treatment A Then Treatment C | Part 2: Treatment B Then Treatment D | Part 2: Treatment D Then Treatment B
Started | 7 | 7 | 0 | 0
Completed | 7 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1: Treatment Period 3
Arm/Group | Part 1: Treatment A Then Treatment B Then Treatment C | Part 1: Treatment B Then Treatment A Then Treatment C | Part 2: Treatment B Then Treatment D | Part 2: Treatment D Then Treatment B
Started | 7 | 7 | 0 | 0
Completed | 7 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2: Treatment Period 1
Arm/Group | Part 1: Treatment A Then Treatment B Then Treatment C | Part 1: Treatment B Then Treatment A Then Treatment C | Part 2: Treatment B Then Treatment D | Part 2: Treatment D Then Treatment B
Started | 0 | 0 | 5 (These are participants which were assigned for that particular treatment/group.) | 6 (These are participants which were assigned for that particular treatment/group.)
Completed | 0 | 0 | 5 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Part 2: Treatment Period 2
Arm/Group | Part 1: Treatment A Then Treatment B Then Treatment C | Part 1: Treatment B Then Treatment A Then Treatment C | Part 2: Treatment B Then Treatment D | Part 2: Treatment D Then Treatment B
Started | 0 | 0 | 5 | 6
Completed | 0 | 0 | 5 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Sisunatovir 200 mg: Participants received treatment A or B or C in any period of Part 1.
- Part 2: Sisunatovir 200 mg: Participants received treatment B or D in any period of Part 2.
- Total: Total of all reporting groups
Arm/Group | Part 1: Sisunatovir 200 mg | Part 2: Sisunatovir 200 mg | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 7 | 5 | 12
  45-64 Years | 6 | 6 | 12
  >=65 Years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 12 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 13 | 8 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 11 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Time Zero to The Time of The Last Quantifiable Concentration (AUClast) of Sisunatovir PIC Versus (vs) WGT in a Fasted State, Part 1
Description: AUClast was calculated using linear/log trapezoidal method. Treatment A = sisunatovir 200 mg PIC under fasted condition; reference treatment. Treatment B = sisunatovir 200 mg WGT under fasted condition; test treatment.
Time Frame: Pre-dose (0 hour), 1, 2, 3, 4, 5, 6, 8, 10,12 hours post-dose on Day 1; 24, 36 hours post-dose on Day 2; 48 hours post-dose on Day 3 of Period 1-3; 72 hours post-dose on Day 4 of period 3
Population: Pharmacokinetic (PK) parameter analysis set included all randomized participants who received at least one dose of study medication and in whom at least 1 plasma PK parameter was calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/ mL)
Groups:
- Part 1: Treatment A: Participants received treatment A on Day 1 of either Period 1 or Period 2.
- Part 1 Treatment B: Participants received treatment B on Day 1 of either Period 1 or Period 2.
Arm/Group | Part 1: Treatment A | Part 1 Treatment B
Number analyzed (Participants) | 14 | 14
nanogram*hour per milliliter (ng*hr/ mL) | 646.6 (97) | 380.5 (123)
Statistical Analysis 1: Comparison: Part 1: Treatment A vs Part 1 Treatment B; Analysis was performed using mixed effect model with sequence, period and treatment as fixed effects and participant within the sequence as a random effect; Test type: Other; Ratio of adjusted geometric means = 58.84, 90% CI 2-sided [40.45 to 85.60] — The ratio (test/reference) and 90% CIs are expressed as percentages. Treatment A = reference; treatment B = test

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUCinf) of Sisunatovir PIC vs WGT in Fasted State, Part 1
Description: AUCinf was calculated as AUClast + (Clast*/kel), where Clast is the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis, and kel is the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve. Treatment A = sisunatovir 200 mg PIC under fasted condition; reference treatment. Treatment B = sisunatovir 200 mg WGT under fasted condition; test treatment.
Time Frame: as for outcome 1
Population: PK parameter analysis set included all randomized participants who received at least one dose of study medication and in whom at least 1 plasma PK parameter was calculated. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram* hour per milliliter (ng*hr/mL)
Arm/Group | Part 1: Treatment A | Part 1 Treatment B
Number analyzed (Participants) | 13 | 13
nanogram* hour per milliliter (ng*hr/mL) | 784.4 (65) | 457.2 (104)
Statistical Analysis 1: Comparison: Part 1: Treatment A vs Part 1 Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means = 56.93, 90% CI 2-sided [38.71 to 83.73] — The ratio (test/reference) and 90% CIs are expressed as percentages. Treatment A = reference; treatment B = test

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Sisunatovir PIC vs WGT in a Fasted State, Part 1
Description: Treatment A = sisunatovir 200 mg PIC under fasted condition; reference treatment. Treatment B = sisunatovir 200 mg WGT under fasted condition; test treatment.
Time Frame: as for outcome 1
Population: PK parameter analysis set included all randomized participants who received at least one dose of study medication and in whom at least 1 plasma PK parameter was calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/ mL)
Arm/Group | Part 1: Treatment A | Part 1 Treatment B
Number analyzed (Participants) | 14 | 14
nanogram per milliliter (ng/ mL) | 63.78 (126) | 31.97 (179)
Statistical Analysis 1: Comparison: Part 1: Treatment A vs Part 1 Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means = 50.13, 90% CI 2-sided [33.01 to 76.13] — The ratio (test/reference) and 90% CIs are expressed as percentages. Treatment A = reference; treatment B = test

4. Secondary Outcome: AUClast of Sisunatovir WGT Under Fasted vs With a High-fat Meal, Part 1
Description: AUClast was calculated using linear/log trapezoidal method. Treatment B = sisunatovir 200 mg WGT under fasted condition; reference treatment. Treatment C = sisunatovir 200 mg WGT with high-fat meal; test treatment.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram* hour per milliliter (ng*hr/mL)
Groups:
- Part 1 Treatment C: Participants received treatment C on Day 1 of Period 3.
Arm/Group | Part 1 Treatment B | Part 1 Treatment C
Number analyzed (Participants) | 14 | 14
nanogram* hour per milliliter (ng*hr/mL) | 380.5 (123) | 770.6 (88)
Statistical Analysis 1: Comparison: Part 1 Treatment B vs Part 1 Treatment C; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means = 202.52, 90% CI 2-sided [138.43 to 296.27] — The ratio (test/reference) and 90% CIs are expressed as percentages. Treatment B = reference; treatment C = test

5. Secondary Outcome: AUCinf of Sisunatovir WGT Under Fasted vs With a High-fat Meal, Part 1
Description: AUCinf was calculated as AUClast + (Clast*/kel), where Clast is the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis, and kel is the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve. Treatment B = sisunatovir 200 mg WGT under fasted condition; reference treatment. Treatment C= sisunatovir 200 mg WGT with high-fat meal; test treatment.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram* hour per milliliter (ng*hr/mL)
Arm/Group | Part 1 Treatment B | Part 1 Treatment C
Number analyzed (Participants) | 13 | 13
nanogram* hour per milliliter (ng*hr/mL) | 457.2 (104) | 896.6 (68)
Statistical Analysis 1: Comparison: Part 1 Treatment B vs Part 1 Treatment C; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means = 196.11, 90% CI 2-sided [131.01 to 293.55] — The ratio (test/reference) and 90% CIs are expressed as percentages. Treatment B = reference; treatment C = test

6. Secondary Outcome: Cmax of Sisunatovir WGT Under Fasted vs With a High-fat Meal, Part 1
Description: Treatment B = sisunatovir 200 mg WGT under fasted condition; reference treatment. Treatment C= sisunatovir 200 mg WGT with high-fat meal; test treatment.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1 Treatment B | Part 1 Treatment C
Number analyzed (Participants) | 14 | 14
nanogram per milliliter (ng/mL) | 31.97 (179) | 73.61 (97)
Statistical Analysis 1: Comparison: Part 1 Treatment B vs Part 1 Treatment C; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means = 230.22, 90% CI 2-sided [145.53 to 364.20] — The ratio (test/reference) and 90% CIs are expressed as percentages. Treatment B = reference; treatment C = test

7. Secondary Outcome: AUClast of Sisunatovir WGT Under Fasted vs With a Low-fat Meal, Part 2
Description: AUClast was calculated using linear/log trapezoidal method. Treatment B = sisunatovir 200 mg WGT under fasted condition; reference treatment. Treatment D= sisunatovir 200 mg WGT with low-fat meal; test treatment.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram* hour per milliliter (ng*hr/mL)
Groups:
- Part 2: Treatment B: Participants received treatment B on Day 1 of either Period 1 or Period 2.
- Part 2 Treatment D: Participants received treatment D on Day 1 of either Period 1 or Period 2.
Arm/Group | Part 2: Treatment B | Part 2 Treatment D
Number analyzed (Participants) | 11 | 11
nanogram* hour per milliliter (ng*hr/mL) | 744.5 (123) | 916.0 (65)
Statistical Analysis 1: Comparison: Part 2: Treatment B vs Part 2 Treatment D; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means = 122.84, 90% CI 2-sided [93.61 to 161.19] — The ratio (test/reference) and 90% CIs are expressed as percentages. Treatment B = reference; treatment D= test

8. Secondary Outcome: AUCinf of Sisunatovir WGT Under Fasted vs With a Low-fat Meal, Part 2
Description: AUCinf was calculated as AUClast + (Clast*/kel), where Clast is the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis, and kel is the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve. Treatment B = sisunatovir 200 mg WGT under fasted condition; reference treatment. Treatment D= sisunatovir 200 mg WGT with low-fat meal; test treatment.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram* hour per milliliter (ng*hr/mL)
Arm/Group | Part 2: Treatment B | Part 2 Treatment D
Number analyzed (Participants) | 10 | 11
nanogram* hour per milliliter (ng*hr/mL) | 996.4 (49) | 957.4 (62)
Statistical Analysis 1: Comparison: Part 2: Treatment B vs Part 2 Treatment D; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means = 104.69, 90% CI 2-sided [94.54 to 115.94] — The ratio (test/reference) and 90% CIs are expressed as percentages. Treatment B = reference; treatment D= test

9. Secondary Outcome: Cmax of Sisunatovir WGT Under Fasted vs With a Low-fat Meal, Part 2
Description: Treatment B = sisunatovir 200 mg WGT under fasted condition; reference treatment. Treatment D= sisunatovir 200 mg WGT with low-fat meal; test treatment.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 2: Treatment B | Part 2 Treatment D
Number analyzed (Participants) | 11 | 11
nanogram per milliliter (ng/mL) | 68.69 (97) | 85.88 (50)
Statistical Analysis 1: Comparison: Part 2: Treatment B vs Part 2 Treatment D; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means = 124.59, 90% CI 2-sided [93.46 to 166.09] — The ratio (test/reference) and 90% CIs are expressed as percentages. Treatment B = reference; treatment D= test

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs): Part 1
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were any AEs that occurred following start of treatment up to 35 days post last dose. Treatment A= sisunatovir 200 mg PIC under fasted condition; treatment B = sisunatovir 200 mg WGT under fasted condition and treatment C= sisunatovir 200 mg WGT with a high-fat meal.
Time Frame: From start of study treatment on Day 1 up to 35 days after last dose of study drug (maximum up to 43 days)
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Treatment B: Participants received treatment B on Day 1 of either Period 1 or Period 2.
Arm/Group | Part 1: Treatment A | Part 1: Treatment B | Part 1 Treatment C
Number analyzed (Participants) | 14 | 14 | 14
Participants | 3 | 6 | 3

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs): Part 2
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were any AEs that occurred following start of treatment up to 35 days post last dose. Treatment B = sisunatovir 200 mg WGT under fasted condition and treatment D= sisunatovir 200 mg WGT with a low-fat meal.
Time Frame: From start of study treatment on Day 1 up to 35 days after last dose of study drug (maximum up to 39 days)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Treatment B: Participants received treatment B on Day 1 of in either Period 1 or Period 2.
- Part 2: Treatment D: Participants received treatment D on Day 1 of in either Period 1 or Period 2.
Arm/Group | Part 2: Treatment B | Part 2: Treatment D
Number analyzed (Participants) | 11 | 11
Participants | 2 | 2

12. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Part 1
Description: Laboratory parameters included: Hematology (Eosinophils/Leukocytes) and Urinalysis (Urine Hemoglobin). Clinically significant laboratory abnormality findings were based on investigator discretion. Clinical significance was determined by the investigator. Treatment A= sisunatovir 200 mg PIC under fasted condition; treatment B = sisunatovir 200 mg WGT under fasted condition and treatment C= sisunatovir 200 mg WGT with a high-fat meal.
Time Frame: From start of study treatment on Day 1 up to 35 days after last dose of study drug (maximum up to 43 days)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 Treatment A: Participants received treatment A on Day 1 of either Period 1 or Period 2.
- Part 1: Treatment B: Participants received treatment B on Day 1 of in either Period 1 or Period 2.
Arm/Group | Part 1 Treatment A | Part 1: Treatment B | Part 1 Treatment C
Number analyzed (Participants) | 14 | 14 | 14
Participants | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Part 2
Description: Laboratory parameters included: Hematology (Eosinophils/Leukocytes) and Urinalysis (Urine Hemoglobin). Clinically significant laboratory abnormality findings were based on investigator discretion. Clinical significance was determined by the investigator. Treatment B = sisunatovir 200 mg WGT under fasted condition and treatment D= sisunatovir 200 mg WGT with a low-fat meal.
Time Frame: From start of study treatment on Day 1 up to 35 days after last dose of study drug (maximum up to 39 days)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment B | Part 2 Treatment D
Number analyzed (Participants) | 11 | 11
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Findings: Part 1
Description: Vital signs (temperature, respiratory rate, pulse, systolic and diastolic blood pressure) were obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Clinically significant vital signs findings were based on investigator discretion. Treatment A= sisunatovir 200 mg PIC under fasted condition; treatment B = sisunatovir 200 mg WGT under fasted condition and treatment C= sisunatovir 200 mg WGT with a high-fat meal.
Time Frame: From start of study treatment on Day 1 up to 35 days after last dose of study drug (maximum up to 43 days)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Treatment A | Part 1: Treatment B | Part 1 Treatment C
Number analyzed (Participants) | 14 | 14 | 14
Participants | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Findings: Part 2
Description: Vital signs (temperature, respiratory rate, pulse, systolic and diastolic blood pressure) were obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Clinically significant vital signs findings were based on investigator discretion. Treatment B = sisunatovir 200 mg WGT under fasted condition and treatment D= sisunatovir 200 mg WGT with a low-fat meal.
Time Frame: From start of study treatment on Day 1 up to 35 days after last dose of study drug (maximum up to 39 days)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment B | Part 2 Treatment D
Number analyzed (Participants) | 11 | 11
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With Clinically Significant 12-lead Electrocardiogram (ECG) Findings: Part 1
Description: A standard 12-lead ECGs utilizing limb leads were collected using an ECG machine that automatically calculated the heart rate (HR) and measures pulse rate (PR), QT, and QTc corrected using Fridericia's formula (QTcF) intervals and QRS complex with the participant in a supine position after at least 5 minutes of rest. Following ECG parameters were analyzed: post-dose QTcF interval is increased by ≥60 ms from the baseline and is >450 ms; or an absolute QT value is ≥500 ms for any scheduled ECG. Clinically significant ECG abnormality findings were based on investigator discretion. Treatment A= sisunatovir 200 mg PIC under fasted condition; treatment B = sisunatovir 200 mg WGT under fasted condition and treatment C= sisunatovir 200 mg WGT with a high-fat meal.
Time Frame: From start of study treatment on Day 1 up to 35 days after last dose of study drug (maximum up to 43 days)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Treatment A | Part 1: Treatment B | Part 1 Treatment C
Number analyzed (Participants) | 14 | 14 | 14
Participants | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Clinically Significant 12-lead Electrocardiogram (ECG) Findings: Part 2
Description: A standard 12-lead ECGs utilizing limb leads were collected using an ECG machine that automatically calculated the heart rate (HR) and measures pulse rate (PR), QT, and QTc corrected using Fridericia's formula (QTcF) intervals and QRS complex with the participant in a supine position after at least 5 minutes of rest. Following ECG parameters were analyzed: post-dose QTcF interval is increased by ≥60 ms from the baseline and is >450 ms; or an absolute QT value is ≥500 ms for any scheduled ECG. Clinically significant ECG abnormality findings were based on investigator discretion. Treatment B = sisunatovir 200 mg WGT under fasted condition and treatment D= sisunatovir 200 mg WGT with a low-fat meal.
Time Frame: From start of study treatment on Day 1 up to 35 days after last dose of study drug (maximum up to 39 days)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment B | Part 2 Treatment D
Number analyzed (Participants) | 11 | 11
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment on Day 1 up to 35 days after last dose of study drug (maximum up to 43 days for Part 1) and (maximum up to 39 days for Part 2)
Groups:
- Part 1 Treatment B; Part 2 Treatment B: Participants received treatment B on Day 1 of in either Period 1 or Period 2.
Arm/Group | Part 1 Treatment A | Part 1 Treatment B | Part 1 Treatment C | Part 2 Treatment B | Part 2 Treatment D
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 3/14 | 6/14 | 3/14 | 2/11 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Treatment A (N=14) | Part 1 Treatment B (N=14) | Part 1 Treatment C (N=14) | Part 2 Treatment B (N=11) | Part 2 Treatment D (N=11)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 2 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT05994963/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT05994963/SAP_001.pdf